CLINICAL TRIAL: NCT07136207
Title: Research on Delirium Recognition in Neurocritical Patients Based on Facial Expression Behavior Patterns
Brief Title: Development and Validation of Delirium Recognition Using Computer Vision in Neuro-critical Patients
Status: Recruiting | Type: Observational
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: Affiliated Jinyang Hospital of Guizhou Medical University (Unknown); Affiliated Hospital of Guizhou Medical University (Unknown)
Responsible Party: Sponsor
Other Study IDs: PX2023021
Record Dates: First submitted 2025-07-18; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Delirium; Artificial Intelligence (AI)
Keywords: Delirium; Artificial Intelligence (AI); neurocritical care units; Facial recognition
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Neurocritical non-delirium patients: For neurocritical non-delirium patients, the investigators record facial expression videos, which are used during model development to compare with the facial expressions of delirium patients.
- Neurocritical delirium patients: The investigators record facial expression videos of neurocritical delirium patients and perform frame sampling on the videos to analyze and extract the facial expression features specific to delirium. Based on this analysis, the investigators develop a model for delirium recognition in neurocritical patients.

SUMMARY:
This research project employs machine learning algorithms integrated with computer vision, image processing, and pattern recognition technologies to perform digital analysis of facial expression behaviors in neurocritical care patients with delirium. By constructing multidimensional high-level features of delirium, the investigators have established a classification model based on behavioral. The primary objective of this study is to address the critical challenge of achieving precise and efficient delirium diagnosis in neurologically critically ill patients through automated facial expression behavior recognition.

DETAILED DESCRIPTION:
This study is a prospective cohort study approved by the Ethics Committee of Beijing Tiantan Hospital. It aims to support the accurate and efficient diagnosis of delirium in neurocritical patients through a facial expression recognition system. A mobile application was developed for this study, collaboratively designed by senior clinicians and engineers from the Institute of Computing Technology, Chinese Academy of Sciences. The application is based on a stimulus paradigm designed using CAM-ICU (Confusion Assessment Method for the Intensive Care Unit) questions to record dynamic facial videos of neurocritical patients following delirium evaluation based on the DSM-V criteria.

Patients were assessed for delirium and facial expression behavior data were collected twice daily during ICU admission, in two time slots: 8:00-10:00 AM and 8:00-10:00 PM, following the study's inclusion and exclusion criteria. A trained and experienced specialist used the gold standard DSM-V to diagnose delirium. Within five minutes after completing the assessment, dynamic facial behavior video data were collected to prepare images for subsequent model development.

Various image preprocessing and data augmentation techniques were employed to prepare the images for the VGG16 model. These techniques are standard for running convolutional neural network (CNN) models. Using the "preprocess_input"function from the Keras VGGFace module, the investigators standardized image color and size to ensure that each image met the expected input requirements for model training. For data augmentation, the investigators applied TensorFlow's "ImageDataGenerator" function to perform horizontal flipping, rotation, scaling, width and height shifting, and shearing. These augmentation techniques created a more diverse dataset, helping to prevent overfitting and improving the model's generalizability to new faces.

The investigators developed a binary classification model to identify delirium using a CNN with a pretrained backbone. The VGG16 model, based on deep learning, was adopted, leveraging transfer learning from VGGFace2, which possesses pre-existing facial feature recognition capabilities. Transfer learning allowed us to utilize prior knowledge to detect features more quickly, accurately, and with lower computational cost. The VGGFace2 model was employed for training.

Model performance was evaluated through internal validation at Beijing Tiantan Hospital and external validation at Guiyang Second People's Hospital, with metrics including accuracy, sensitivity, specificity, and F1 score. Additionally, to address the "black box" issue of machine learning, occlusion heatmap techniques were used to identify the most critical facial regions for delirium assessment, with the results visualized on a virtual face.

This model aims to support precise and efficient identification of delirium in neurocritical care units.

ELIGIBILITY:
Inclusion Criteria:

1. Neurocritical patients admitted to the ICU, including postoperative neurosurgical patients, stroke patients, and those receiving ICU care due to other neurological conditions.
2. Age over 18 years.
3. Signed informed consent.

Exclusion Criteria:

1. Age under 18 years.
2. Persistent coma (GCS ≤ 8) within 7 days pre- and post-surgery, making delirium assessment impossible.
3. Did not survive more than 24 hours in the ICU.
4. Patients with facial paralysis, post-traumatic facial disfigurement, or other conditions that could significantly affect facial recognition.
5. Exclusion of patients with severe dementia, Parkinson's disease, depression, or other conditions that might impact facial emotional expressions.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study selects neurocritical patients as the population and collects facial expression data from both delirium and non-delirium patients.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-08-30 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Accuracy of the delirium prediction model | Through study completion, an average of 1 year
  The accuracy of the delirium prediction model will be calculated as the proportion of correct predictions among total predictions.
Sensitivity of the delirium prediction model | Through study completion, an average of 1 year
  Sensitivity (true positive rate) will be assessed as the proportion of actual delirium cases correctly identified by the model.
Specificity of the delirium prediction model | Through study completion, an average of 1 year
  Specificity (true negative rate) will be calculated as the proportion of non-delirium cases correctly identified by the model.

SECONDARY OUTCOMES:
F1 Score of the delirium prediction model | Through study completion, an average of 1 year
  The F1 score, the harmonic mean of precision and recall, will be used to evaluate the balance between sensitivity and specificity.
AUC of the facial feature curve for delirium patients | Through study completion, an average of 1 year
  The area under the curve (AUC) of the receiver operating characteristic (ROC) curve derived from facial features will be used to assess the discriminatory performance of the model.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
This study involves collecting facial information of patients, which pertains to their privacy. To protect participants' confidentiality, all data will be uniformly destroyed after the study is completed. The investigators will not share or disclose patients' information to other researchers.

REFERENCES:
- [Background] Heintz TA, Badathala A, Wooten A, Cu CW, Wallace A, Pham B, Wallace AW, Cobert J. Preliminary Development and Validation of Automated Nociception Recognition Using Computer Vision in Perioperative Patients. Anesthesiology. 2025 Apr 1;142(4):726-737. doi: 10.1097/ALN.0000000000005370. Epub 2025 Jan 13. PMID 39804295
- [Background] Atee M, Hoti K, Parsons R, Hughes JD. A novel pain assessment tool incorporating automated facial analysis: interrater reliability in advanced dementia. Clin Interv Aging. 2018 Jul 16;13:1245-1258. doi: 10.2147/CIA.S168024. eCollection 2018. PMID 30038491
- [Background] Goldberg TE, Chen C, Wang Y, Jung E, Swanson A, Ing C, Garcia PS, Whittington RA, Moitra V. Association of Delirium With Long-term Cognitive Decline: A Meta-analysis. JAMA Neurol. 2020 Nov 1;77(11):1373-1381. doi: 10.1001/jamaneurol.2020.2273. PMID 32658246
- [Background] Aldecoa C, Bettelli G, Bilotta F, Sanders RD, Audisio R, Borozdina A, Cherubini A, Jones C, Kehlet H, MacLullich A, Radtke F, Riese F, Slooter AJ, Veyckemans F, Kramer S, Neuner B, Weiss B, Spies CD. European Society of Anaesthesiology evidence-based and consensus-based guideline on postoperative delirium. Eur J Anaesthesiol. 2017 Apr;34(4):192-214. doi: 10.1097/EJA.0000000000000594. PMID 28187050
- [Background] Ely EW, Margolin R, Francis J, May L, Truman B, Dittus R, Speroff T, Gautam S, Bernard GR, Inouye SK. Evaluation of delirium in critically ill patients: validation of the Confusion Assessment Method for the Intensive Care Unit (CAM-ICU). Crit Care Med. 2001 Jul;29(7):1370-9. doi: 10.1097/00003246-200107000-00012. PMID 11445689
- [Background] Ahmed A, Garcia-Agundez A, Petrovic I, Radaei F, Fife J, Zhou J, Karas H, Moody S, Drake J, Jones RN, Eickhoff C, Reznik ME. Delirium detection using wearable sensors and machine learning in patients with intracerebral hemorrhage. Front Neurol. 2023 Jun 9;14:1135472. doi: 10.3389/fneur.2023.1135472. eCollection 2023. PMID 37360342
- [Background] Al-Hindawi A, Vizcaychipi M, Demiris Y. A Dual-Camera Eye-Tracking Platform for Rapid Real-Time Diagnosis of Acute Delirium: A Pilot Study. IEEE J Transl Eng Health Med. 2024 May 7;12:488-498. doi: 10.1109/JTEHM.2024.3397737. eCollection 2024. PMID 39050621
- [Background] Oh J, Cho D, Park J, Na SH, Kim J, Heo J, Shin CS, Kim JJ, Park JY, Lee B. Prediction and early detection of delirium in the intensive care unit by using heart rate variability and machine learning. Physiol Meas. 2018 Mar 27;39(3):035004. doi: 10.1088/1361-6579/aaab07. PMID 29376502
- [Background] Eeles E, Tronstad O, Teodorczuk A, Flaws D, Fraser JF, Dissanayaka N. Face and content validity of a mobile delirium screening tool adapted for use in the medical setting (eDIS-MED): Welcome to the machine. Australas J Ageing. 2024 Jun;43(2):415-419. doi: 10.1111/ajag.13288. Epub 2024 Feb 28. PMID 38415380
- [Background] Nejati V, Khorrami AS, Fonoudi M. Neuromodulation of facial emotion recognition in health and disease: A systematic review. Neurophysiol Clin. 2022 Jun;52(3):183-201. doi: 10.1016/j.neucli.2022.03.005. Epub 2022 Apr 12. PMID 35428551

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-09-26): https://cdn.clinicaltrials.gov/large-docs/07/NCT07136207/Prot_SAP_000.pdf
  • Informed Consent Form (2024-09-26): https://cdn.clinicaltrials.gov/large-docs/07/NCT07136207/ICF_001.pdf